CLINICAL TRIAL: NCT05231174
Title: Efficacy of Using Large Language Model to Assist in Diabetic Retinopathy Detection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yingfeng Zheng, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022KYPJ258
Record Dates: First submitted 2022-01-29; First posted 2022-02-09 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Diagnosis; Diabetic Retinopathy
MeSH Terms: conditions — Disease; Diabetic Retinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A self-evlaution tool based on Large Language Model (Experimental): The self-evlaution tool, powered by a large language model, processes user queries through a comprehensive generation, decision, action, and safety framework to deliver optimal responses. The system's key features include retrieval-augmented in-context learning, which enhances the responses generated by sourcing information from reliable websites. It also incorporates a Guardrail module to mitigate potential harmful content in the responses by validating the content before delivery. Additionally, the system features a Self-checking memory module that maintains essential clinical characteristics across multi-turn dialogues, ensuring consistent and continuous interactions with users.
  Interventions: Other: A self-evlaution tool based on Large Language Model

INTERVENTIONS:
Other: A self-evlaution tool based on Large Language Model — Following the baseline assessment, participants will be guided to use a self-evaluation tool independently to assess their risk of diabetic retinopathy (DR). This tool is a fusion of a conversational AI system based on LLM and an existing logistic diagnostic model.
  The AI system is designed to collect clinical variables, including age, duration of diabetes, Body Mass Index (BMI), and insulin usage. Additionally, clinical test data such as mean arterial pressure, HbA1c, serum creatinine, and microalbuminuria will be extracted from a local dataset using the patient's name and ID. Once collected, these data will be transmitted to a server-based diagnostic model for further analysis to determine the presence of DR.

SUMMARY:
With the increase in population and the rising prevalence of various diseases, the workload of disease diagnosis has sharply increased. The accessibility of healthcare services and long waiting times have become common issues in the public health medical system, with many primary patients having to wait for extended periods to receive medical services. There is an urgent need for rapid, accurate, and low-cost diagnostic services.

ELIGIBILITY:
Inclusion Criteria The study will include adults aged 18 years and above who have been diagnosed with Type 2 diabetes but have not previously been screened for DR. Participants must demonstrate good compliance with clinical examinations, and provide informed consent.

Exclusion criteria The study will exclude patients who have previously been diagnosed with DR, those who have recently undergone eye surgery, and those with other significant eye diseases that could potentially confound the results of DR screening. Individuals with ocular, auditory, or cognitive impairments that prevent the use of mobile phones or reading will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 535 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
AUROC of the self-evaluation tool | Immediately after using the chatbot
  The performance of the self-evaluation tool is evaluated with accuracy with reference to the diagnostic labels by senior ophthalmologists based on fundus photos.

CONTACTS AND LOCATIONS:
Overall Officials: Yingfeng Zheng, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhognshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No